CLINICAL TRIAL: NCT06651749
Title: Hemodynamic Effects of a High Dose Versus Low Dose Propofol During Induction of Anesthesia. a Randomized Comparative Trial.
Brief Title: Hemodynamic Effects of a High Dose Versus Low Dose Propofol During Induction of Anesthesia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MS332/2024
Record Dates: First submitted 2024-10-19; First posted 2024-10-22 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-05

CONDITIONS: Hemodynamic Effects of Propofol
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high dose propofol during induction of anesthesia. (Active Comparator): this group will be given high dose propofol 2.5mg/kg during induction of anesthesia.
  Interventions: Drug: Propofol injection
- low dose propofol during induction of anesthesia. (Active Comparator): this group will be given low dose propofol 1.5mg/kg during induction of anesthesia.
  Interventions: Drug: Propofol injection

INTERVENTIONS:
Drug: Propofol injection — hemodynamic changes of a high dose versus low dose propofol during induction of anesthesia.

SUMMARY:
The investigators will test the hemodynamic effects of a high dose versus low dose Propofol during induction of anesthesia.

DETAILED DESCRIPTION:
A. Preoperative settings:

In the anesthesia clinic, an informed written consent will be obtained from every patient one day before the surgery. All patients will be assessed preoperatively by careful history taking full physical examination, and laboratory evaluation.

B. Intraoperative settings:

On the arrival to operation room; standard ASA monitors will be attached automatic blood pressure measurements, five-lead ECG monitor, capnography and finger pulse oximetry will be applied, The baseline value was measured.

Measurement of mean arterial blood pressure by non-invasive blood pressure monitoring(NIBP) at selected time interval would be obtained as follows:

* baseline value( NIBP "systolic, diastolic and mean value" and HR): 1 minute pre-injection
* 1 minute post injection
* 3 minutes post injection
* 5 minutes post injection
* Final value :7 minutes post injection

The investigators will calculate the percentage difference of lowest mean arterial blood pressure from baseline value using the following formula:

(Baseline mean blood pressure - lowest value mean blood pressure)/ Baseline mean blood pressure

* An intravenous infusion of ringer acetate 3ml/kg will be started.
* Pre-oxygenation with 100% O2 on 8 L/min for 3 min via face mask will be started.
* Induction of anesthesia would be done by using propofol dosage according to the group

  1. Group LDP will receive 1.5mg/kg propofol during induction of anesthesia.
  2. Group HDP will receive 2.5mg/kg propofol during induction of anesthesia.
* In group LDP, if the patient is still showing signs of awareness or intact eyelash reflex within two minutes post injection, the investigators will add 1mg/kg propofol and the patient will be shifted to the HDP group.
* Fentanyl would be given during induction 2mic/kg IV.
* Atracurium besylate 0.5 mg/kg IV will be given to facilitate tracheal intubation, and anaesthesia will be maintained with 1 to 1.5% isoflurane.
* After orotracheal intubation, mechanical ventilation will be started, controlled mechanical ventilation will be achieved by tidal volumes of 8-10 mL/Kg and frequency of ventilation of up to 12-14 breaths/min to maintain normocapnia: end-tidal pressure CO2 (ET CO2) at the level of 35 ± 5 mm Hg and Positive End Expiratory Pressure (PEEP) of 5-10 cm H2O.
* Supplemental boluses of Atracurium besylate 0.1 mg/kg IV will be administered every 20 minutes to maintain muscle relaxation during surgery. Anaesthesia will be maintained with isoflurane 1-1.5% to maintain the HR and MAP within 20% of pre-induction values and/or Heart Rate (HR) < 85 beats/ min during surgical stimulation.
* Regular automated monitoring : NIBP "systolic, diastolic and mean value" and HR /5minutes
* At the end of the surgery, each patient will be extubated upon meeting the extubation criteria.
* Intraoperatively, any increase or decrease of HR, hypotension or hypertension will be managed as required.
* If the patient sustains Bradycardia (defined as: HR ≤50 bpm for 3 minutes), atropine 0.6 mg/kg increments will be administered till acceptable response.
* If the patient sustains Hypotension (defined as a decrease in systolic blood pressure >20%-30% of baseline value for 3 minutes), administration of ephedrine5-6 mg increments, and fast intravenous fluid bolus (250 ml crystalloids).
* If the patient sustains Hypertension (defined as an increase in systolic blood pressure >20%-30% of baseline value for 3 minutes ), raising the end-tidal isoflurane concentration to 2% and 0.5 μg/kg IV bolus of fentanyl will be administered till acceptable response after exclusion of causes other than sympathetic response to surgical stimulus .
* The whole study period will be attended and supervised by the most skilled person in the study group.

  c.Postoperative settings: The patients will be transferred to the post-anaesthesia care unit and will be put under observation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: from 21 years old till 40 years old.
2. Patients with ASA classification I and II.
3. Undergoing a scheduled elective surgery.

Exclusion Criteria:

1. Declining to give written informed consent.
2. ASA classification III-V.
3. Patients with class III (morbid) obesity or more (BMI >40 Kg/m2)
4. Patients with severe intraoperative hypotension requiring large volume of intravascular fluid treatment.
5. Severe or uncontrolled hypertension (NIBP> 150/100) , congestive heart failure, moderate to severe valvular heart disease , uncontrolled arrhythmia , heart rate>100bpm .
6. Significant hepatic or renal disorder.
7. Patients with uncontrolled diabetes mellitus type 1 or type 2(evidenced by autonomic dysfunction or organ complications, ischemic heart disease or cerebrovascular disease).
8. Patients who were pregnant (positive pregnancy test) or menstruating.
9. Anemia with hemoglobin level <9.0 g/dL
10. Hypersensitivity to soybean oil, egg lecithin, or glycerol.
11. Medical substance abuse.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage difference of lowest mean arterial blood pressure from baseline value. | from injection till 7 minutes post-injection
  will

CONTACTS AND LOCATIONS:
Overall Officials: Hadeer S Saied, M.B.B.CH, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams university, Cairo, Abbaseya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data will be shared once study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: before may 2025
Access Criteria: free